CLINICAL TRIAL: NCT03970616
Title: A Phase 1b/2, Open-Label, Study of Tivozanib in Combination With Durvalumab in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Tivozanib in Combination With Durvalumab in Subjects With Advanced Hepatocellular Carcinoma
Acronym: DEDUCTIVE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to regulatory approval of newer therapeutic options and slower than anticipated accrual.
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-18-121
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tivozanib; durvalumab

STUDY DESIGN:
Intervention Model Description: Phase 1 followed by expansion cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tivozanib in Combination with Durvalumab (Experimental): Tivozanib in Combination with Durvalumab
  Interventions: Drug: Tivozanib; Drug: Durvalumab

INTERVENTIONS:
Drug: Tivozanib — Dose level 1: 1.0mg for 21 days followed by 7 days rest; Dose level -1: 1.0mg every other day
  Other Names: Fotivda
Drug: Durvalumab — 1500mg every 28 days
  Other Names: Imfinzi

SUMMARY:
This study will evaluate the safety, tolerability, DLTs, MTD, and preliminary anti tumor activity of tivozanib in combination with durvalumab in subjects with advanced HCC.

ELIGIBILITY:
Subjects to be included

1. ≥ 18 years old
2. Signed and dated written informed consent
3. Histologically or cytologically or radiologically confirmed unresectable locally advanced or metastatic hepatocellular carcinoma. Measurable or evaluable disease by RECIST 1.1 criteria. Patients can be either untreated or have progressed on both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor.

   o Patients who may have progressed on bevacizumab and atezolizumab who have any suggestion of pseudo-progression, should remain on bevacizumab and atezolizumab until progression is confirmed.
4. Child-Pugh Class A.
5. ECOG performance status ≤ 1 (see Appendix A) and life expectancy ≥ 3 months.
6. Body weight > 30 kg
7. Measured creatinine clearance (crCL) >40 mL/min or calculated crCL >40 mL/min as determined by Cockcroft-Gault (using actual body weight) Males CrCL = Weight (kg) × (140 - Age) 72 × serum creatinine (mg/dL) Females CrCL = Weight (kg) × (140 - Age) 85 × serum creatinine (mg/dL)
8. Sexually active pre-menopausal female subjects (and female partners of male subjects) must use highly effective contraceptive measures, while on study and for at least 90 days after the last dose of study drug. Sexually active male subjects must use adequate contraceptive measures, while on study and for at least 90 days after the last dose of study drug. All fertile male and female subjects and their partners must agree to use a highly effective method of contraception.

Note - COVID-19 testing is not required prior to enrollment into the protocol, however, institutional guidelines on testing should be followed.

Subjects to be excluded

1. Subjects who have received prior systemic treatment for HCC except for both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor.
2. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of study drug.
3. Brain metastases or spinal cord compression. Subjects with suspected brain metastases at screening should have an MRI (preferred) or CT scan each preferable with IV contrast of the brain prior to study entry. Brain metastases will not be recorded on RECIST Target Lesions at baseline.
4. Any of the following hematologic abnormalities:

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) < 1500 per mm3
   * Platelet count < 75,000 per mm3
5. Any of the following serum chemistry or urinalysis abnormalities:

   * Total bilirubin > 2 × ULN (>2.5 mg/dL in subjects with Gilbert's syndrome)
   * AST or ALT > 5 × ULN
   * Alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis)
   * Serum creatinine > 1.5 × ULN •> 2+ proteinuria
6. History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy (eg, no lactulose, rifaximin, etc if used for purposes of hepatic encephalopathy).
7. GI Bleeding (eg, esophageal varices or ulcer bleeding) within 12 months. (Note: For patients with a history of GI bleeding for more than 12 months or assessed as high risk for esophageal variceal bleed by the Investigator, adequate endoscopic therapy according to institutional standards is required).
8. Clinically meaningful ascites defined as ascites requiring non-pharmacologic intervention (eg, paracentesis) to maintain symptomatic control, within 6 months prior to the first scheduled dose. Subjects on stable doses of diuretics for ascites for ≥ 2 months are eligible.
9. Main portal vein thrombosis (Vp4) as documented on imaging. (VP4 is defined as portal vein thrombosis in the main trunk of the portal vein or a portal vein branch contralateral to the primarily involved lobe (or both).
10. For subjects who require ongoing therapeutic anti-coagulation or anti-platelet therapy; the subject must be off either therapy for at least 7 days prior to the first dose of investigational product. Low-dose aspirin for cardiac prophylaxis/protection is permitted per local institutional standards.
11. Patients co-infected with HBV and HCV. HBV positive [presence of hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10IU/ml)]; HCV positive (presence of anti-HCV antibodies).
12. Major surgery (as defined by the investigator) within 28 days prior to first dose of IP or still recovering from prior surgery. Local procedures (eg, core needle biopsy, and prostate biopsy) are allowed if completed at least 3 days prior to the administration of the first dose of study treatment.
13. Significant cardiovascular disease, including:

    * Clinically symptomatic heart failure. Subjects with a history of heart failure must have an ECHO or MUGA scan to document left ventricular ejection fraction (LVEF) > 45% prior to start of protocol therapy
    * Any New York Heart Association classification ≥ Class 2 (prefer Class 0 or 1)
    * Any stenting procedure within the last 3 months
    * Venous thromboembolism or arterial thromboembolism within the last 3 months
    * Any IVC tumor thrombosis
    * History of a hemorrhagic event (i.e., GI bleed within 6 months)
    * Uncontrolled hypertension: blood pressure >150/95 mmHg on more than 2 antihypertensive medications, on two consecutive measurements obtained at least 24 hours apart. Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 2 weeks prior to start of protocol therapy.
    * Myocardial infarction within 3 months prior to start of protocol therapy
14. Subjects with delayed healing of wounds, ulcers, and/or bone fractures
15. Serious/active infection or infection requiring parenteral antibiotics
16. Inadequate recovery from any prior surgical procedure; major surgical procedure within 4 weeks prior to start of protocol therapy.
17. Inability to comply with protocol requirements
18. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study drug and low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer of lentigo maligna without evidence of disease
19. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
20. Patients with a history or current HBV infection (detectable HBV DNA), should be placed on anti-viral treatment and tested at every cycle for HBV DNA viral load.
21. Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation or to more than 30% of the bone marrow within 4 weeks before the first dose of study intervention.
22. Treatment with systemic hormonal therapy within 3 weeks prior to start of protocol therapy, with the exception of:

    * Hormonal therapy for appetite stimulation or contraception
    * Nasal, ophthalmic, inhaled and topical steroid preparations
    * Oral replacement therapy for adrenal insufficiency
    * Low-dose maintenance steroid therapy (equivalent of prednisone 10mg/day) for other conditions
    * Hormone replacement therapy such as testosterone
23. Strong CYP3A4 inducers (see Appendix B) within 2 weeks prior to start of, or during, protocol therapy.
24. Prior exposure to tivozanib or durvalumab. For subjects who have received prior atezolizumab:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a Grade ≥ 3 immune-related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy. Note: Participants with an endocrine AE of Grade ≤ 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
25. History of allogeneic organ transplantation
26. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Subjects with vitiligo or alopecia
    * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Subjects without active disease in the last 5 years may be included but only after consultation with Medical Monitor
    * Subjects with celiac disease controlled by diet alone
27. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent
28. History of leptomeningeal carcinomatosis
29. History of active primary immunodeficiency
30. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
31. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
32. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study
33. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving study drug and up to 30 days after the last dose of study drug.
34. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
35. Previous study drug assignment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Approximately 24 months; Through study completion
  To establish the safety of tivozanib in combination with durvalumab in subjects with untreated advanced hepatocellular carcinoma (HCC).
Incidence of Treatment Emergent Adverse Events (TEAEs) | Approximately 24 months; Through study completion
  To establish the safety of tivozanib in combination with durvalumab in subjects with advanced hepatocellular carcinoma (HCC) previously treated with both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor in a prior line of therapy.

SECONDARY OUTCOMES:
Response Rate (Objective Response Rate) | Approximately 24 months
  To estimate the response rate of tivozanib in combination with durvalumab in subjects with untreated advanced HCC.
Progression Free Survival (PFS) | Approximately 24 months
  To estimate the progression free survival (PFS) of tivozanib in combination with durvalumab in subjects with untreated advanced HCC.
Overall Survival (OS) | Approximately 24 months; Through study completion
  To estimate the overall survival (OS) of tivozanib in combination with durvalumab in subjects with untreated advanced HCC.
Response Rate (Objective Response Rate) | Approximately 24 months
  To estimate the response rate of tivozanib in combination with durvalumab in subjects with advanced HCC previously treated with both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor in a prior line of therapy.
Progression Free Survival (PFS) | Approximately 24 months; Through study completion
  To estimate the progression free survival (PFS) of tivozanib in combination with durvalumab in subjects with advanced HCC previously treated with both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor in a prior line of therapy.
Overall Survival (OS) | Approximately 24 months; Through study completion
  To estimate the overall survival (OS) of tivozanib in combination with durvalumab in subjects with advanced HCC previously treated with both bevacizumab and atezolizumab or both bevacizumab and atezolizumab in combination with a second immune checkpoint inhibitor in a prior line of therapy.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - University of California - Irvine, Orange, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston (UTHealth), Houston, Texas
  - The University of Texas Health Science Center at Tyler (UTHealth), Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmood S, Li D, Lee A, Rowe J, Beg M, Kasturi V, Iyer R, Abrams T, Dayyani F. A multicenter, phase Ib/II, open-label study of tivozanib with durvalumab in advanced hepatocellular carcinoma (DEDUCTIVE). Future Oncol. 2022 Dec;18(40):4465-4471. doi: 10.2217/fon-2022-0844. Epub 2023 Mar 13. PMID 36912078